CLINICAL TRIAL: NCT02601677
Title: Deep Brain Stimulation of Nucleus Accumbens/Anterior Limb of Internal Capsule to Prevent Treatment-Refractory Obsessive Compulsive Disorder
Brief Title: Deep Brain Stimulation of NAc/ALIC to Prevent Treatment-Refractory Obsessive Compulsive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Principal Investigator, Guodong Gao, Neurosurgery Department, Tang-Du Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OCD-DBS
Record Dates: First submitted 2015-11-08; First posted 2015-11-10 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Obsessive Compulsive Disorder
Keywords: Obsessive Compulsive Disorder; Deep Brain Stimulation; Nucleus accumbens
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Deep Brain Stimulation; Fluoxetine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Deep Brain Stimulation (Experimental): Continuous deep brain stimulation of bilateral nucleus accumbens
  Interventions: Procedure: Deep brain stimulation
- Standard Control (Active Comparator): Fluoxetine
  Interventions: Drug: Fluoxetine

INTERVENTIONS:
Procedure: Deep brain stimulation — Deep brain stimulation of bilateral Nucleus accumbens/Anterior Limb of Internal Capsule
  Arms: Deep Brain Stimulation
Drug: Fluoxetine — Fluoxetine is one of selective serotonin reuptake inhibitors(SSRIs).
  Arms: Standard Control

SUMMARY:
Nucleus accumbens/anterior limb of internal capsule play important roles in the process of treatment-refractory obsessive compulsive disorder, deep brain stimulation of nucleus accumbens/anterior limb of internal capsule will inhibit its activity and thus to effectively prevent the disorder.

DETAILED DESCRIPTION:
Obsessive-compulsive disorder (OCD) is characterized by obsessions (persistent thoughts) and compulsions (repetitive ritualistic behaviour). Core symptoms of OCD cause remarkable distress and often perceived as inappropriate. The prevalence of OCD in the general population is estimated between 1% and 3%. It is a psychiatric illness that can lead to chronic functional impairment. Treatment options for OCD include cognitive behavioural therapy (CBT) and/or pharmacotherapy. Even when the best treatment options are used, approximately 10% of these patients remain severely affected and are considered therapy-refractory resulting in marked suffering and impairment in self-care, work and social life. More recently, deep brain stimulation (DBS) has been investigated as a therapy for refractory OCD, and the procedure was granted a limited humanitarian device exemption by the FDA in 2009. For these patients, deep brain stimulation (DBS), a neurosurgical treatment that involves stereotactic implantation of electrodes in specific deep-seated brain regions, has emerged as a new treatment option.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of OCD following the diagnostic and statistical manual of mental disorders-fourth edition (DSM-IV) criteria for OCD;
2. Duration of illness: min. 5 year;
3. 18 years old <Age <60 years old;
4. Severe form of OCD, as evidenced by: a score≥25 on the Y-BOCS, a score > 4 on the CGI scale, a score≤40 on the GAF ("global assessment of functioning).
5. All patients were lack of response to drug therapy after adequate administration (defined as more than 12 weeks at the maximum tolerated dose) of at least four different medications, lack of response to CBT (Cognitive Behaviour Therapy)over the course of 1 year of therapy or after 20 sessions.
6. Normal cognitive status and ability to understand and comply with instructions for multiple therapies.
7. Good overall health.

Exclusion Criteria:

1. Present or past history of psychotic symptoms.
2. Severe personality disorders;
3. Any clinically significant neurological disorder or medical illnesses affect ;
4. brain function, other than motor tics or Gilles de la Tourette syndrome;
5. Patient currently treated with anticoagulant or antiplatelet drug;
6. Patient with contraindication for surgery or anesthesia;
7. Inability to undergo awaked operation;
8. Infection, coagulopathy, significant cardiac or other medical risk factors for surgery;
9. Patient with contraindication for MRI scanning (cardiac pacemaker, pregnancy, metal in body, severe claustrophobia), abnormal brain MRI or serious inter current disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-11; Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | 6 month

SECONDARY OUTCOMES:
Clinical Global Impression (CGI) | 6 month
Global assessment of functioning (GAF) | 6 month
The Hamilton Anxiety Scale (HAM-A) | 6 month
The Hamilton Rating Scale for Depression (HAM-D) | 6 month
Sheehan Disability Scale (SDS) | 6 month
Event related potentials(ERPs) | Baseline,3 month,6 month and 12 month
local field potential(LFP) | in surgery,7 days after surgery
Change in two static positron emission tomography(PET) images study | Baseline and 6month follow-up